CLINICAL TRIAL: NCT07348952
Title: Different Transcutaneous Electrical Nerve Stimulation Modes in Pudendal Neuralgia Post-prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Tawfik, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mohamed-Phd
Record Dates: First submitted 2026-01-01; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Pudendal Neuralgia; Post Prostatectomy
MeSH Terms: conditions — Pudendal Neuralgia | interventions — Transcutaneous Electric Nerve Stimulation; Gabapentin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional Transcutaneous Electrical Nerve Stimulation (Experimental): was composed of 30 patients who received the conventional transcutaneous electrical nerve stimulation in addition to the traditional physical therapy and medical care for 3 months.
  Interventions: Device: conventional Transcutaneous Electrical Nerve Stimulation; Other: Traditional physical therapy; Drug: Gabapentin
- Acupuncture-like) transcutaneous Electrical Nerve Stimulation (Active Comparator): that was composed of 30 patients who received the SLR (Acupuncture-like) transcutaneous Electrical Nerve Stimulation in addition to the traditional physical therapy and medical care for 3 months
  Interventions: Device: Acupuncture-like) transcutaneous Electrical Nerve Stimulation; Other: Traditional physical therapy; Drug: Gabapentin

INTERVENTIONS:
Device: conventional Transcutaneous Electrical Nerve Stimulation — A Transcutaneous Electrical Nerve Stimulation stimulator Zimmer Elektromedizingalva 5, from Germany was used. The Transcutaneous Electrical Nerve Stimulation treatment will be applied once daily, three times per week for three months. Each session lasts 20 minutes, using two electrodes over the perineal area on the Centrum tendineum and two under the buttocks at the ischial spines. The patient will be in a comfortable supine hook-lying position with abducted hips. The electrode surface area must be at least 4 cm² to prevent burns, and the interelectrode distance will not be less than the electrode's diameter. Adhesive electrodes will be used, or alternatively, moistened with jelly and secured with adhesive tape in the recommended areas. Square wave form with a frequency of 80-100 Hz and intensity of 10-30 milli ampere, associated with a pulse width of 50-60 µsec, generates comfortable paresthesia (tingling) without significant muscle contractions or fasciculations.
  Arms: conventional Transcutaneous Electrical Nerve Stimulation
Device: Acupuncture-like) transcutaneous Electrical Nerve Stimulation — A Transcutaneous Electrical Nerve Stimulation stimulator Zimmer Elektromedizingalva 5, from Germany was used. The Transcutaneous Electrical Nerve Stimulation treatment will be applied once daily, three times per week for three months. Each session lasts 20 minutes, using two electrodes over the perineal area on the Centrum tendineum and two under the buttocks at the ischial spines. The patient will be in a comfortable supine hook-lying position with abducted hips. The electrode surface area must be at least 4 cm² to prevent burns, and the interelectrode distance will not be less than the electrode's diameter. Adhesive electrodes will be used, or alternatively, moistened with jelly and secured with adhesive tape in the recommended areas. Square wave form with a frequency under 10 Hz and an intensity of 30 to 80 milli ampere will produce rhythmic, visible muscle contractions lasting 300-400 msec, tailored to the subject's tolerance at the same electrode placement.
  Arms: Acupuncture-like) transcutaneous Electrical Nerve Stimulation
Other: Traditional physical therapy — Traditional physical therapy for pudendal neuralgia following prostatectomy emphasizes conservative pain management and restoring pelvic floor function. This includes patient education, activity modification, postural correction, and supportive cushions to reduce perineal pressure. Pain relief methods involve thermal applications and relaxation techniques, while pelvic floor therapy focuses on muscle relaxation through manual therapy and myofascial release. Treatment introduces gentle stretching, neural mobilization, and stabilization exercises, tailored to the patient's needs and often coordinated with a multidisciplinary team.
Drug: Gabapentin — First-line treatments for neuropathic pain include gabapentin, pregabalin, tricyclic antidepressants (like amitriptyline), and SNRIs (such as duloxetine). NSAIDs and simple analgesics may address associated inflammatory pain but are less effective for neuropathic pain specifically. Muscle relaxants can help with pelvic floor spasms, and topical agents like lidocaine offer localized relief. For persistent symptoms, pudendal nerve blocks may be performed by specialists.

SUMMARY:
The purpose of this study was to evaluate the therapeutic efficacy of two different Transcutaneous Electrical Nerve Stimulation modes in improving the pudendal neuralgia and its intractable perineal pain.

DETAILED DESCRIPTION:
The need for this study will be developed from the lack in quantitative knowledge and information in the published studies about the effects of two different transcutaneous electrical nerve stimulation modes in cases of pudendal neuralgia. The significance of this study will be raised from the persistence of this neuralgia and its intractable pain that may result in severe morbidity with repeated local injections, pain medications and numerous surgical attempts to alleviate pain as well as the increase in the period of hospitalization plus the delay in returning to normal life. So, this study will be conducted to add new information about the effect of different transcutaneous electrical nerve stimulation modes in relieving chronic pudendal neuralgia post-prostatectomy, which may help the field of physical therapy and patients suffering from pudendal neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be chosen after a routine medical examination.
* All patients will be approximately the same age (from 50-60 years old).
* All patients have chronic pudendal neuralgia post-prostatectomy surgery.
* They have not take another physical therapy electro- modality except the traditional physical therapy in the form of pelvic floor exercises.
* All of them will be non smokers and will be under own prescribed medications described by their physicians.
* The pain is located in the pudendal nerve distribution area.
* Pain intensity increased in the sitting position.
* There were no symptoms of nocturnal pain.
* Pain with no objective sensory impairment.
* Pain was relieved by diagnostic pudendal nerve block.
* Another clinical standard provides extra support to the diagnosis of pudendal neuralgia.
* Pain symptoms may be associated with sexual dysfunction.

Exclusion Criteria:

* Patients have simple tailbone, gluteus muscle or lower abdominal pain, or only paroxysmal pain, or only pruritic symptoms, and/or having imaging anomalies that may explain the symptoms.
* Patients who take anticoagulant drugs or have any coagulation disorder.
* Patients who will be unable to complete the study.
* Patients with pain, which is caused by malignant or autoimmune diseases.
* Patients with life threatening disorders as renal failure, myocardial infarction or others will be excluded from the study.
* Patients who suffering from skin diseases, diabetes, varicose veins, trauma and peripheral vascular diseases will be excluded.
* Patients who suffering from myasthenia gravis, hyperthyroidism, hemorrhage, acute viral diseases, acute tuberculosis, mental disorders or those with pace makers will be excluded from the study

Ages: 50 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * All patients will be approximately the same age (from 50-60 years old).
  * All patients have chronic pudendal neuralgia post-prostatectomy surgery
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
measurement of Serum cortisol level | at baseline and 12 weeks
  Normal morning serum cortisol levels range from 9 to 25 µg/dL, and patients with painful conditions tend to exhibit higher-than-normal serum cortisol levels. Estimation of serum cortisol levels will be performed before and after 3 months of the treatment program. A venous blood sample (8 cubic centimeter) will be collected in the morning, centrifuged, and stored at -20 °C until analysis.

SECONDARY OUTCOMES:
assessment of pain intensity | at baseline and 12 weeks
  Pain intensity was evaluated using the Visual Analog Scale (VAS), which features a 10-cm line marked from no pain (0) to worst imaginable pain (10). Participants indicated their pain level on this line, and the distance from the zero point was recorded as the pain score. VAS assessments occurred before and after treatment and are recognized as a valid and reliable method for quantifying pain intensity in clinical research.
assessment of the carbamazepine intake | at baseline and 12 weeks
  it will be used to evaluate the improvement in the chronic pudendal neuralgia post-prostatectomy and its intractable perineal pain

CONTACTS AND LOCATIONS:
Locations (1):
- out-clinics of the general surgery department in Om-El Misrieen hospital, Giza, Egypt